CLINICAL TRIAL: NCT07375433
Title: Heart Failure With Preserved Ejection Fraction in Patients With Сhronic Obstructive Pulmonary Disease: Clinical Course and Prognosis
Acronym: HIPSTER
Status: Recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Kazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 06-08/25
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Heart Failure With Preserved Ejection Fraction (HFpEF; Diagnosis)
Keywords: Heart failure; Heart failure with Preserved Ejection Fraction; Biomarkers; COPD; Prognosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease; Heart Failure | interventions — Echocardiography; Spirometry; Plethysmography, Whole Body; Walk Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Сhronic Obstructive Pulmonary Disease: Patients hospitalized with a verified diagnosis of COPD. Patients with a confirmed diagnosis in accordance with instrumental and clinical criteria.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Spirometry; Diagnostic Test: Body plethysmography; Diagnostic Test: 6-Minute Walk Test (6MWT); Diagnostic Test: laboratory biomarker analysis

INTERVENTIONS:
Diagnostic Test: Echocardiography — Transthoracic echocardiography at rest: with determination of epicardial fat tissue thickness, epicardial adipose tissue thickness (EAT), E/e', interventricular septum thickness, left ventricular posterior wall thickness, and end-diastolic dimension
Diagnostic Test: Spirometry — Spirometry is the most common of the pulmonary function tests, which measures the lung capacity and airway patency (volume and speed of air) during quiet and forced breathing.
Diagnostic Test: Body plethysmography — Body plethysmography is a non-invasive lung function test performed in a sealed booth (body box) that measures total lung volume, functional residual capacity, and airway resistance by using Boyle's Law to track pressure and volume changes as a patient breathes, providing crucial data for diagnosing conditions like COPD and asthma, and differentiating them from other lung disorders
Diagnostic Test: 6-Minute Walk Test (6MWT) — The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity
Diagnostic Test: laboratory biomarker analysis — Routine and special laboratory tests

SUMMARY:
Study aim is comparison of heart failire with preserved ejection fraction (HFpEF) detection rate in patients with Сhronic Obstructive Pulmonary Disease (COPD) and the clinical course and prognosis in patients with COPD depending on HFpEF presence.

DETAILED DESCRIPTION:
Study aim of Investigation "Heart Failure with Preserved Ejection Fraction in Patients with Сhronic Obstructive Pulmonary Disease: Clinical Course and Prognosis" (HIPSTER) is comparison of heart failire with preserved ejection fraction (HFpEF) detection rate in patients with Сhronic Obstructive Pulmonary Disease (COPD) and the clinical course and prognosis in patients with COPD depending on HFpEF presence.

It is assumed that newly diagnosed HFpEF will occur in at least 6% (COPD PRIORITY data) of cases, and, the presence of HFpEF will negatively affect both the manifestations of the disease and the outcomes and prognosis

During the study it is planned to:

1. Perform a retrospective analysis of patient records, determine the frequency of intracardiac hemodynamic disorders, corresponding with the criteria for HFpEF and compare them with the diagnosis in clinical records.
2. Identify the patients with previously undiagnosed HFpEF among patients with COPD, and evaluate the frequency of cardiorespiratory comorbidity.
3. Examine the general clinical and biochemical blood test parameters in the study groups (as part of a routine in-patient examination).
4. Evaluate echocardiography parameters in the study groups (as part of a routine protocol + epicardial adipose tissue thickness (EAT), E/e', interventricular septum thickness, left ventricular posterior wall thickness, and end-diastolic dimension (EDD).
5. Compare spirometry and body plethysmography parameters in the groups depending on the presence of HFpEF criteria.
6. Compare the functional status (Six-Minute Walk Test, 6MWT) in the study groups.
7. Evaluate patient's vital status after 12 months, information about hospitalizations and their reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Verified diagnosis of COPD;
2. Patients hospitalized with COPD;
3. Citizenship of the Russian Federation;
4. Patients aged 50 to 70 years;
5. Patient consent to participate in the study.

Exclusion Criteria:

1. Lack of Russian Federaion citizenship;
2. Patient's refusal to participate in the study;
3. Any chronic diseases, other than COPD, that affect the prognosis, in the acute and/or decompensated stage;
4. Mental disorders.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Generic russian population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary composite endpoin | 1 year
  Primary composite endpoint: all-cause death, rehospitalizations, major adverse cardiovascular events (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Olga D Dzhioeva, MD, associate professor, Study Director — National Medical Research Center for Therapy and Preventive Medicine; Diana I Abdulganieva, MD, professor, Study Director — Kazan State Medical University
Locations (2):
- Russia (2):
  - Kazan State Medical University, Kazan'
  - National Medical Research Center for Therapy and Preventive Medicine, Moscow

IPD SHARING:
Plan to Share IPD: Undecided